CLINICAL TRIAL: NCT03735524
Title: The Inflammatory Synaptopathy as a Target of Exercise Therapy in the Fight Against Multiple Sclerosis
Brief Title: Exercise-based Therapy for Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neuromed IRCCS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NeuromedIRCCS
Record Dates: First submitted 2018-10-10; First posted 2018-11-08 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-11

CONDITIONS: Multiple Sclerosis
Keywords: exercise, synaptopathy, inflammation
MeSH Terms: conditions — Multiple Sclerosis; Motor Activity; Inflammation | interventions — Exercise; Rehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Conventional rehabilitation
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Different exercises will be adopted including: repetition of different movements for ambulation and stair climbing, repetition of crossed patterns of movements for coordination, postural reactions while standing with eyes open and closed and oscillatory boards for balance, strengthening lower limb muscles, and low-intensity and long-duration static stretching of iliopsoas, rectus femoris, hamstrings, triceps surae, and lumbar spinal muscles for muscular flexibility and range of motion. In addition, advanced robotic therapy will be used to standardize rehabilitative treatment and to obtain more objective indexes of motor function. The Lokomat exoskeleton and the Biodex stability system will be used.
  Other Names: Rehabilitation

SUMMARY:
Exercise is reported to have significant beneficial effects in Multiple Sclerosis (MS) patients, particularly with respect to cardiovascular function, aerobic capacity, muscular strength and ambulatory performance. Inflammation-mediated synaptic alterations have been measured by means of transcranial magnetic stimulation (TMS) and found to correlate with disability level in MS. Due to their plastic nature, synapses represent a good therapeutic target that is sensitive to environmental stimulation, such as physical exercise.

The aim of this study is to evaluate the effect of exercise in reducing peripheral inflammation that drives the synaptic pathology and neurodegeneration occurring in the brain of MS patients. Recruited patients will be given a therapeutic exercise program, consisting of 3 hours of treatment per day, 6 days/week for 4 weeks. The program will be applied on hospitalised patients to ensure adherence to the program and reducing the risk of abandonment. The rehabilitation program will be planned by a physician specialised in physical and rehabilitation medicine and will consist of both passive and active therapeutic exercises specifically aimed at restoring or maintaining muscular flexibility, range of motion, balance, coordination of movements, postural passages and transfers, and ambulation. The day of recruitment (t0) patients will undergo radiological and neurological examination. The effect of exercise will be evaluated with respect to neurologic function, mood and neurophysiological parameters, autonomic system function, and peripheral marker levels assessed at t0 and after 4 weeks (t1). A second time point will be included (t2, 8 weeks after the end of the treatment) to address long-term effects, with analysis limited to neurologic and mood measurements and peripheral marker levels.

DETAILED DESCRIPTION:
Clinical manifestations of Multiple Sclerosis (MS) indicate the involvement of motor, sensory, visual, and autonomic systems as well as brain circuits implicated in cognition and emotion.

Due to the complexity and the heterogeneity of the disease course and the clinical symptoms, the search for the appropriate personalized treatment and the disease management remains a challenging issue. Nowadays, it is increasingly recognized that MS treatment and care demand a multi-disciplinary approach, including non-pharmacological interventions, aimed to improve quality of life (QoL) and engagement in daily-life activities. Active-rehabilitation or exercise is currently considered as the form of non-medical interventions that best meets these requirements.

In the context of MS, there is now general agreement on the positive effects of exercise for both relapsing remitting (RR) and progressive (P) MS patients. Significant effects have been described for cardiovascular functions, aerobic capacity, muscular strength and ambulatory performance. Even if clear conclusions cannot be drawn, other outcomes, like balance and depression seem to be positively influenced by exercise. Symptoms linked to autonomic dysfunction caused by sympathovagal imbalance, like altered heart rate variability (HRV) and correlating with the load of inflammation in MS may benefit from exercise, being the physical activity an important modulator of the peripheral nervous system. However, the DMT potential of exercise is still overlooked, since only few studies have investigated the influence of exercise on inflammation and neurodegeneration, the main pathogenic events in MS with unclear and, to some extent, contrasting data.

This longitudinal study aims is designed to enrol at least 35 MS patients to perform a conventional 4 weeks rehabilitation program. Physical therapy will be performed for 6 days/week for 4 weeks and will consist of 3 hours of treatment. The rehabilitation program will be planned by a physician specialized in physical and rehabilitation medicine and will consist of both passive and active therapeutic exercises specifically aimed at restoring or maintaining muscular flexibility, range of motion, balance, coordination of movements, postural passages and transfers, and ambulation. According to the patient's disability status, different therapeutic exercises will be performed by qualified physiotherapists. Moreover, intensity of exercise will be tailored to the level of patient's disability. To avoid fatigue and to increase patient's tolerance to the exercises, compensative pauses will be included. Moreover, genotype analysis from peripheral blood cells will be performed to identify single nucleotide polymorphisms (SNPs) in coding regions and/or gene regulators (microRNA or proteins) involved in MS synaptic transmission alterations, like NGF, PDGF, which might correlate to clinical parameters described as both primary and secondary outcomes.

Statistical analysis will be performed by IBM SPSS Statistics 15.0. Data will be tested for normality distribution through the Kolmogorov-Smirnov test. Differences between pre- and post-values will be analyzed using parametric Student's t-test for matched pairs, or if necessary, nonparametric Wilcoxon signed-rank test for matched pairs. Changes in categorical variables will be assessed by McNemar test. Correlation analysis will be performed by calculating Pearson or Spearman coefficients as appropriate. Data will be presented as the mean (standard deviation, sd) or median (25th- 75th percentile). The significance level is established at p<0.05.

Sample size calculation was performed according to the following criteria. Supposing that in MS patients the cytokine values in particular the TNF levels after exercise therapy decrease in a manner similar to that showed in the study by Hedegaard et al (2008), the investigators can estimate that the therapy will have a medium effect on TNF values, d=0.59, calculating a pre-mean value equal to 2611.2 (standard deviation, sd=1586.96) and post-exercise equal to 1249.1 (sd=1261.89), a correlation between pre-post values equals to -0.326. To detect as significant a moderate effect with a power of 95%, assuming a two-sided a=0.05 and applying a Wilcoxon signed-rank test for matched pairs, the investigators estimate a total number of 35 patients. The analysis was performed by G*POWER v3.1.9.2.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent to the study;
* Diagnosis of MS definite according to 2010 revised McDonald's criteria (Polman et al., 2011);
* Age range 18-65 (included);
* EDSS range between 4,5 and 6,5 (included);
* Ability to participate to the study protocol.

Exclusion Criteria:

* Inability to provide written informed consent to the study;
* Altered blood count;
* Female with positive pregnancy test at baseline or having active pregnancy plans in the following months after the beginning of the protocol;
* Contraindications to gadolinium (MRI);
* Contraindications to TMS;
* Patients with comorbidities for neurological disease other than MS, included other neurodegenerative chronic diseases or chronic infections (i.e tubercolosis, infectious hepatitis, HIV/AIDS);
* Unstable medical condition or infections;
* Use of medications with increased risk of seizures (i.e. Fampridine, 4-Aminopyridine);
* Concomitant use of drugs that may alter synaptic transmission and plasticity (cannabinoids, L-dopa, antiepiletics, nicotine, baclofen, SSRI, botulinum toxin).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2019-05 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Changes in clinical disability (EDSS) | Changes from baseline (time 0, t0), 4 weeks after the end of exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Clinical severity will be measured by the expanded disability status scale (EDSS): the EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Changes in clinical disability: Multiple Sclerosis Functional Composite (MSFC) | Changes from baseline (time 0, t0), 4 weeks after the end of exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  The Multiple Sclerosis Functional Composite (MSFC) is a three-part composite clinical measure. Three variables were recommended as primary measures: Timed 25-Foot walk; 9-Hole Peg Test; and Paced Auditory Serial Addition Test (PASAT-3"). The results from each of these three tests are transformed into Z-scores and averaged to yield a composite score for each patient at each time point.
  There are 3 components:
  1. the average scores from the four trials on the 9-HPT;
  2. the average scores of two 25-Foot Timed Walk trials;
  3. the number correct from the PASAT-3. The scores for these three dimensions are combined to create a single score that can be used to detect change over time. This is done by creating Z-scores for each component.
  MSFC Score = {Zarm, average + Zleg, average + Zcognitive} / 3.0 (Where Zxxx =Z-score) Increased scores represent deterioration in the 9-HPT and the 25-Foot Timed Walk, whereas decreased scores represent deterioration in the PASAT-3.
Changes in clinical disability (VA) | Changes from baseline (time 0, t0), 4 weeks after the end of exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  The best corrected visual acuity (VA) that will performed in a well-lit room using Snellen and low-contrast letter acuity (LCLA) charts to assess clinical severity.

SECONDARY OUTCOMES:
Changes in Mood-depressive trait | Changes from baseline (time 0, t0) to the end of the 4-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Depression will be assessed by means of the Beck Depression Inventory-Second Edition (BDI-II) (Watson et al, 2014).
Changes in Mood-anxiety trait | Changes from baseline (time 0, t0) to the end of the 4-week exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Anxiety will be assessed by State-Trait Anxiety Inventory (STAI) form Y (STAI-Y), a 40-item self-administered questionnaire measuring anxiety as a state (situational anxiety) or trait (long-standing proneness to anxious situations).
Neurophysiological assessment | Changes from baseline (time 0, t0) to the end of the 4-week exercise protocol (time 1, t1)
  Cortical excitability will be probed with transcranial magnetic stimulation (TMS) using Magstim devices (The Magstim Company, Whitland, Dyfed, UK). One stimulator will be connected to a figure-of-eight coil (external wing diameter 70 mm) placed tangentially over the scalp in the optimal position for eliciting motor evoked potentials (MEPs) in the first dorsal interosseous (FDI) muscle of the dominant hand. To test the interhemispheric inhibition (IHI) we will apply a paired-pulse (conditioning-test) TMS paradigm. Paired pulses will be given with interstimulus intervals (ISIs) of 10 and 40 ms. LTP will be assessed by the intermittent theta-burst stimulation (iTBS) protocol. iTBS consists of three-pulse bursts given at 80% AMT and 50 Hz frequency, repeated every 200 ms (i.e. at 5 Hz) and delivered over the FDI muscle hot spot, for a total number of 600 stimuli. We will record and average fifteen MEPs of about 1 mV peak-to-peak in amplitude at baseline before iTBS.
Changes in autonomic function | Changes from baseline (time 0, t0) to the end of the 4-week exercise protocol (time 1, t1)
  Heart rate variability (HRV) will be assessed under standardized environmental conditions. ECG will be recorded by standard methods. The analysis will be performed in the frequency domain using a dedicated software. Stable heart rate (HR) periods of 5 minutes duration will be chosen in the last 6 minutes of a 30-minute supine rest. Power spectral analysis will consider a high frequency (HF) component, reflecting mostly vagal activity, and a low frequency (LF) component, reflecting mostly sympathetic activity. Spectral components in normalized units (LFnu, HFnu) will be considered. As an index of sympathovagal balance, we will use the LF/HF ratio.
Changes in peripheral cytokine levels | Changes from baseline (time 0, t0) to the end of 4 week-exercise protocol (time 1, t1) and 8 weeks after the end of exercise protocol (time 2, t2)
  Within few hours after the withdrawal, the peripheral blood will be processed to isolate plasma, serum and cells.
  Peripheral Blood Mononuclear Cells (PBMCs) will be isolated by Ficoll hystopaque gradient centrifugation, according to standard techniques and soon frozen in -80 and next processed to isolate T cells by magnetic immunosorting with FITC-CD3 antibody and microbeads-conjugated anti-FITC antibody (Miltenyi, Biotec). TNF and IL-1b released by T cells in culture medium will be measured by using commercial ELISA kit. Data will be expressed as picograms per milliliter (pg/ml).

CONTACTS AND LOCATIONS:
Overall Officials: Diego Centonze, MD, Principal Investigator — IRCCS Neuromed
Locations (1):
- IRCCS Neuromed, Pozzilli, Isernia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Charron S, McKay KA, Tremlett H. Physical activity and disability outcomes in multiple sclerosis: A systematic review (2011-2016). Mult Scler Relat Disord. 2018 Feb;20:169-177. doi: 10.1016/j.msard.2018.01.021. Epub 2018 Feb 2. PMID 29414293
- [Background] Compston A, Coles A. Multiple sclerosis. Lancet. 2002 Apr 6;359(9313):1221-31. doi: 10.1016/S0140-6736(02)08220-X. PMID 11955556
- [Background] Dalgas U, Stenager E, Jakobsen J, Petersen T, Hansen HJ, Knudsen C, Overgaard K, Ingemann-Hansen T. Resistance training improves muscle strength and functional capacity in multiple sclerosis. Neurology. 2009 Nov 3;73(18):1478-84. doi: 10.1212/WNL.0b013e3181bf98b4. PMID 19884575
- [Background] Deckx N, Wens I, Nuyts AH, Hens N, De Winter BY, Koppen G, Goossens H, Van Damme P, Berneman ZN, Eijnde BO, Cools N. 12 Weeks of Combined Endurance and Resistance Training Reduces Innate Markers of Inflammation in a Randomized Controlled Clinical Trial in Patients with Multiple Sclerosis. Mediators Inflamm. 2016;2016:6789276. doi: 10.1155/2016/6789276. Epub 2016 Jan 20. PMID 26903712
- [Background] Edwards T, Pilutti LA. The effect of exercise training in adults with multiple sclerosis with severe mobility disability: A systematic review and future research directions. Mult Scler Relat Disord. 2017 Aug;16:31-39. doi: 10.1016/j.msard.2017.06.003. Epub 2017 Jun 12. PMID 28755682
- [Background] Feinstein A, DeLuca J, Baune BT, Filippi M, Lassman H. Cognitive and neuropsychiatric disease manifestations in MS. Mult Scler Relat Disord. 2013 Jan;2(1):4-12. doi: 10.1016/j.msard.2012.08.001. Epub 2012 Sep 25. PMID 25877449
- [Background] Feys P, Giovannoni G, Dijsselbloem N, Centonze D, Eelen P, Lykke Andersen S. The importance of a multi-disciplinary perspective and patient activation programmes in MS management. Mult Scler. 2016 Aug;22(2 Suppl):34-46. doi: 10.1177/1352458516650741. PMID 27465614
- [Background] Golzari Z, Shabkhiz F, Soudi S, Kordi MR, Hashemi SM. Combined exercise training reduces IFN-gamma and IL-17 levels in the plasma and the supernatant of peripheral blood mononuclear cells in women with multiple sclerosis. Int Immunopharmacol. 2010 Nov;10(11):1415-9. doi: 10.1016/j.intimp.2010.08.008. Epub 2010 Aug 24. PMID 20797460
- [Background] Motl RW, Sandroff BM, Kwakkel G, Dalgas U, Feinstein A, Heesen C, Feys P, Thompson AJ. Exercise in patients with multiple sclerosis. Lancet Neurol. 2017 Oct;16(10):848-856. doi: 10.1016/S1474-4422(17)30281-8. Epub 2017 Sep 12. PMID 28920890
- [Background] Rampello A, Franceschini M, Piepoli M, Antenucci R, Lenti G, Olivieri D, Chetta A. Effect of aerobic training on walking capacity and maximal exercise tolerance in patients with multiple sclerosis: a randomized crossover controlled study. Phys Ther. 2007 May;87(5):545-55. doi: 10.2522/ptj.20060085. Epub 2007 Apr 3. PMID 17405806
- [Background] Schulz KH, Gold SM, Witte J, Bartsch K, Lang UE, Hellweg R, Reer R, Braumann KM, Heesen C. Impact of aerobic training on immune-endocrine parameters, neurotrophic factors, quality of life and coordinative function in multiple sclerosis. J Neurol Sci. 2004 Oct 15;225(1-2):11-8. doi: 10.1016/j.jns.2004.06.009. PMID 15465080
- [Background] Sternberg Z. Promoting sympathovagal balance in multiple sclerosis; pharmacological, non-pharmacological, and surgical strategies. Autoimmun Rev. 2016 Feb;15(2):113-23. doi: 10.1016/j.autrev.2015.04.012. Epub 2015 May 3. PMID 25945428
- [Background] Studer V, Rocchi C, Motta C, Lauretti B, Perugini J, Brambilla L, Pareja-Gutierrez L, Camera G, Barbieri FR, Marfia GA, Centonze D, Rossi S. Heart rate variability is differentially altered in multiple sclerosis: implications for acute, worsening and progressive disability. Mult Scler J Exp Transl Clin. 2017 Apr 5;3(2):2055217317701317. doi: 10.1177/2055217317701317. eCollection 2017 Apr-Jun. PMID 28607756
- [Background] van den Berg M, Dawes H, Wade DT, Newman M, Burridge J, Izadi H, Sackley CM. Treadmill training for individuals with multiple sclerosis: a pilot randomised trial. J Neurol Neurosurg Psychiatry. 2006 Apr;77(4):531-3. doi: 10.1136/jnnp.2005.064410. PMID 16543538